CLINICAL TRIAL: NCT06591156
Title: Treatment of Miller Class I Gingival Recessions by CAF with or Without Platelet-Rich Fibrin: a Randomized Clinical Controlled Trial
Brief Title: Gingival Recessions Treated by CAF with or Without PRF
Acronym: GR with PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Salgado de Oliveira (Other)
Collaborators: University of Salamanca (Other); A.T. Still University of Health Sciences (Other)
Responsible Party: Principal Investigator, Gustavo Fernandes, DDS, MSc, PhD, PhD, Universidade Salgado de Oliveira
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCP 2020-123
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gingival Recession, Plastic Surgery; Platelet
Keywords: Gingival recession; Platelet-Rich Fibrin; Root coverage; Periodontal plastic surgery
MeSH Terms: conditions — Gingival Recession | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Procedure with PRF membranes (Experimental): Root coverage procedure. One group received PRF membranes.
  Interventions: Procedure: Root coverage
- Control group (Active Comparator): Coronally advanced flap only without any graft or biomaterial
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: Root coverage — Treatment of gingival recession, Miller's Class I or Cairo's RT1, which is the most predictable group to receive interventions without any impairment or problem for the patients.
  After local anesthesia, a horizontal incision was made, delimitating the coronal part of the flap. This horizontal incision of the envelope flap consists of an oblique submarginal incision in the interdental areas that creates a surgical papilla. The incisions continue with the intrasulcular incision in the recession defects and are extended to form an envelope flap between the central and molar. This design facilitates the planned coronal repositioning of the flap tissue on the exposed root surfaces.
  The apical gingival tissue at root exposures is raised to a full thickness to provide the critical part of the flap for root coverage with more thickness. Finally, the most apical portion of the flap is elevated in a split-thickness to facilitate coronal displacement of the flap.
  Other Names: Gingival recession
  Arms: Procedure with PRF membranes
Procedure: control group — Coronally advanced flap without any graft or biomaterial
  Other Names: Control
  Arms: Control group

SUMMARY:
The objective of this study was to compare the efficacy of Coronal Advanced Flap (CAF) alone versus CAF combined with Leukocyte-Platelet-Rich Fibrin (L-PRF) to achieve root coverage in patients with gingival recession. This was assessed by measuring the percentage of root coverage at six months post-surgery. By focusing on the root coverage level, the study aimed to determine whether adding L-PRF to CAF significantly improved over using CAF alone.

The other objective was to provide a comprehensive assessment of the outcomes related to root coverage and overall patient satisfaction. Moreover, different outcomes of recession coverage were assessed, including the percentage of complete root coverage and mean root coverage. These evaluations were intended to offer a more detailed understanding of the possible success of each surgical technique. Additionally, the difference in gingival tissue thickness between the two groups was attempted to measure at six months post-surgery to determine whether the addition of L-PRF to CAF improved tissue quality and stability.

The study also aimed to determine the overall volume gain in gingival tissue in the specific area of recession covered by both techniques, providing information on their regenerative capabilities and the three-dimensional changes in tissue structure.

Furthermore, it sought to analyze the healing and recovery processes by comparing postoperative complications, patient discomfort, and overall recovery time between the two groups. Finally, another goal was to investigate the patient's satisfaction with the aesthetic and functional outcomes of the procedures, evaluating their perceptions of the success of treatment and the quality of life after surgery. This comprehensive approach was designed to ensure that all relevant outcomes were considered, offering a robust evaluation of the effectiveness and benefits of combining CAF with L-PRF and providing comparability with previous and future studies.

The positive hypothesis raised was: CAF combined with L-PRF will: (a) result in significantly greater root coverage compared to CAF alone at six months post-surgery; (b) lead to thicker gingival tissue and better tissue quality compared to CAF alone; (c) will have a faster healing and recovery, with fewer complications in the CAF with L-PRF group compared to the CAF alone group; (d) will report higher satisfaction levels with the treatment outcomes compared to those undergoing CAF alone.

DETAILED DESCRIPTION:
A clinician not involved with the care of participants assessed eligibility and filled out the data form, and after receiving the allocation information from the randomization unit, the surgeon, a clinician not involved in data collection, started the protocolized procedure.

BLOOD COLLECTION: If a patient was assigned to the test group (L-PRF), a designed nurse proceeded to the blood collection to obtain L-PRF. A vein (basilica, cephalic, or median), usually on the inside of the elbow or the back of the hand, was the source of blood. The area where the puncture occurred was cleaned with an antiseptic. An elastic band or pressure cuff was wrapped around the forearm to squeeze the vein and make it more noticeable under the band. This helped the needle find the vein more easily.

As soon as that was done, a needle was placed in the vein, and blood was collected in a clean and sealed plastic tube (Intra Spin™ - Intra-Lock), between 4 and 6 tubes, without anticoagulant. During the process, the band was removed to allow blood to flow normally, and after the blood was collected, the needle was removed, and the puncture site was covered to prevent bleeding. The L-PRF membranes were prepared according to the technique described by Choukroun et al. (2001). Tubes were centrifuged immediately at 2700 rpm for 12 minutes on the centrifugation machine (Intraspin™, Intra-lock®, Florida, USA).

After centrifugation, the gelatinous portion obtained from each tube was removed and separated from the red part with tweezers. The membranes obtained were placed on a sterile metal surface.

The light metal plate and cover of the compression box (e.g., Xpression™ Intra-Lock, Boca Raton, FL, USA) were used to gently compress the L-PRF clots by gravity. After five minutes, the L-PRF membranes could be used.

A protocol of 2700RPM for 12 minutes (RCF-clot = 408g) was used to produce L-PRF membranes with leukocytes and platelets. L-PRF membranes were produced utilizing an Intraspin™ centrifugation device (33° rotor angulation, 50mm radius at the clot, 80mm at the max, Intra-Lock, Boca Raton, Florida, USA) utilizing 9mL glass-coated plastic tubes (Intra-Lock).

SURGICAL PROCEDURE: In case of CEJ undetectable or with 'step,' CEJ restoration was performed prior to the surgical procedure and digital scan (T0).

The coronally advanced flap (CAF) technique for multiple gingival recessions, as described by de Sanctis and Zucchelli, is a minimally invasive surgical procedure with intrasulcular incisions around the affected teeth and horizontal incisions in the interdental areas, preserving the papillae. A split-full-split thickness envelope flap is then elevated, with split-thickness dissection in the papillae and beyond the mucogingival junction and full-thickness at the recession level. This technique avoids vertical releasing incisions, contributing to better blood supply, improved esthetics, and a more comfortable postoperative experience for the patient.

SURGICAL STEP BY STEP: The anesthetic was applied to the intervened area, and a coronal advance flap was created. After local anesthesia, a horizontal incision was made, delimitating the coronal part of the flap. This horizontal incision of the envelope flap consists of an oblique submarginal incision in the interdental areas that creates a surgical papilla. The incisions continue with the intrasulcular incision in the recession defects and are extended to form an envelope flap between the central and molar. This design facilitates the planned coronal repositioning of the flap tissue on the exposed root surfaces.

The envelope flap is raised with a split-full-split approach in the coronal-apical direction, and the oblique interdental incisions are performed, keeping the blade parallel to the long axis of the teeth to dissect the surgical papilla in a split-thickness manner.

The apical gingival tissue at root exposures is raised to a full thickness to provide the critical part of the flap for root coverage with more thickness. Finally, the most apical portion of the flap is elevated in a split-thickness to facilitate coronal displacement of the flap. At the limit of the flap (central and molar), a hemi-utilization was performed to ensure the release of tension and better mobilization of the flap at extremities.

Then, a sharp dissection was performed in the mucosa of the vestibular lining to eliminate muscle tension. It must be considered that the "adequate" coronal displacement of the flap results from eliminating muscle and lip tensions in the apical part of the flap. This way, the flap design incorporates a wide base to ensure adequate blood supply, with the base of the flap being wider than the coronal portion to promote better vascularization and healing. The flap's length should be sufficient to cover the recession defects fully and extend coronally beyond the CEJ of the involved teeth, ensuring complete coverage of the exposed roots and promoting optimal healing.

The epithelium is removed from the anatomical papillae to allow them to fit the surgical papillae at the time of suture. Then, root cleaning is performed with manual Mini-Gracey curettes (LM®, Finland).

In the CAF+L-PRF group, ideal 6 (minimum 4) L-PRF membranes (with dimensions of receptor bed) are fixed together, with resorbable suture six zeros (Novosyn®, BBraun, Melsungen, Germany) and adapted to the root surface at CEJ level with the face of the inner membrane towards the recession.

The flap is then repositioned. Each surgical papilla that was dislocated surgically (concerning the anatomic papilla by the oblique submarginal interdental incisions) is now placed over the de-epithelialized papilla, promoting a rotation of the flap toward the canine and in a coronal direction. One of the key factors for recession coverage techniques is ensuring that the flap can be advanced coronally without any tension. So, if considered necessary, when verifying the reposition of the flap, additional partial-thickness dissection was performed apically to relieve tension and allow for proper positioning of the flap before suture.

After repositioning the flap, it was stabilized with a suspended suture. Sling sutures with 6/0 PTFE (Elasyn®, BBraun, Melsungen, Germany) were used to precisely adapt the buccal flap on the exposed root surfaces and stabilize every surgical papilla.

To ensure standardization of the technique and less variability, the flap was always performed from central to first molar (no vertical incisions), even if there was no recession at the lateral or central level.

ELIGIBILITY:
Inclusion criteria:

* People over 18 years of age
* Nonsmokers or smokers with less than ten cigarettes (self-reported)
* No medical pathology that prevents the application of treatments affects the response of these and the healing process: protein and vitamin deficiency, therapeutic radiation, metabolic disorders (diabetes, hypercalcemia, and others.), drug disorders (antimetabolic, immunosuppressive) and hormonal, allergy to some component of the treatments applied in the study.
* Not be pregnant.
* The presence of oral health with the plaque control record (PCR) and bleeding on probing (BOP)is less than 25%
* At least, the presence of two or more neighboring, or not, gingival recessions Miller class 1 in the anterior upper jaw (central and lateral incisors, canine, first and second premolars.

Exclusion criteria:

* not accepted participation in the study
* not signed the informed consent
* recession greater than Miller's class1 or RT-1
* presence of any non-controlled disease. 4) Gingival recessions present a minimal amount (>1,5 mm) of keratinized tissue (KT) apical to the recession area.

  5) Pocket depth (PD) </=3 mm and CAL interproximal </ = 0 6) Absence of carious lesions, occlusal trauma, or previous root cover procedures.

  7) Absence of a prosthetic crown on experimental teeth.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
PERCENTAGE (%) OF ROOT COVERAGE (PRC) | 6 months
  The primary outcome of this trial was the percentage of root coverage achieved at six months post-surgery. This outcome was chosen due to its high clinical relevance and direct impact on patient care. Clinically, the percentage of root coverage is a crucial measure of success in periodontal surgical procedures aimed at treating gingival recession. It indicates how effectively the exposed root surface has been covered by gingival tissue.
  The objective is to evaluate whether L-PRF, combined with the coronal advancement flap for root coverage in Miller Class 1 recessions in upper front teeth, will show any significant clinical difference in the root coverage percentage compared to the coronal advancement flap alone. We used two methods to measure the percentual of root coverage: one based on the changes in recession depth (standard), and one based on the changes in recession area for comparison.
  This metric represents the exact p
COMPLETE AND MEAN ROOT COVERAGE | 6 months
  % of complete root coverage (%CRC) Complete root coverage indicates that the gingival margin has been successfully repositioned to cover the previously exposed root surface, which is often the primary goal of these treatments. Provides a clear binary outcome (complete vs. incomplete), making it easy to interpret. This measurement is directly correlated with patient satisfaction. Patients typically seek treatment for gingival recession to address aesthetic and sensitivity issues. Patients may only be satisfied when they achieve total coverage of the root surface.
  Mean Root coverage (MRC) This metric represents the average root coverage achieved in a sample or study group, expressed in absolute terms (e.g., millimeters). It is an absolute measurement that provides information about the amount of root coverage achieved, which can be clinically important.

SECONDARY OUTCOMES:
KERATINIZED TISSUE WIDTH GAIN | 6 months
  The gain of keratinized tissue (KTW) is a critical outcome in periodontal surgical procedures aimed at recession coverage due to its substantial impact on periodontal health, treatment stability, and patient satisfaction. Keratinized tissue, characterized by its dense and fibrous nature, plays a crucial role in maintaining gingival health and function. Keratinized tissue provides a more robust barrier against mechanical trauma from brushing and chewing, as well as bacterial invasion. This variable was obtained by a difference in keratinized width at T0 and keratinized tissue width at 6 months. The measurements were obtained by digital measurement.
THICKNESS GAIN | 6 months
  The gain of gingival tissue thickness (GT) is crucial in periodontal surgical procedures aimed at root coverage due to its significant impact on the long-term stability of the gingival tissues, patient comfort, and aesthetic outcomes. Thicker gingival tissues enhance the stability and resilience of the gingival margin, reducing susceptibility to mechanical trauma and bacterial invasion, thus preventing future recession and ensuring the longevity of treatment outcomes.
  These metrics were obtained by superimposing presurgical and postoperative digital models and posterior 3D comparison, as will be discussed in the material and methods.
PAIN AND HEALING ASSESSMENT | 6 months
  An examination of existing wound healing scales in oral surgery shows that they have low use, and their structure does not match the stages of the wound healing process. Because of that, we intend to use a recently proposed novel scale: the IPR (I = inflammatory, P = proliferative, R = remodeling) wound healing scale. This newer scale, already used in implant dentistry, is better for clinical research to evaluate new products that can affect wound healing results. Pain is subjectively assessed by the patient and all other parameters are evaluated by an oral surgeon who is not the operating surgeon.
  The inflammatory phase has the most significant weight in the final score because its impairment can jeopardize the entire series of biological events that lead to early wound healing. The remodeling phase carries the lowest weight because it can spread over several years and involves maintaining a biological balance between matrix degradation and formation which occurs after wound closure.
SUBJECTIVE EVALUATION OF RESULTS BY THE PATIENT | 6 months
  A way to measure the quality of care and the effectiveness of root coverage procedures from the patient's point of view is to use PROMs (patient-reported outcome measures). PROMs are questionnaires that ask the patient about their health status, experience, satisfaction, and expectations before and after treatment. Using PROMS, clinicians can understand the patient's needs, preferences, and values and assess the effect of their interventions on oral health and quality of life. PROMS can also help improve clinician and patient communication and increase shared decision-making and patient participation in their care. There is a discrepancy between how the clinician and the patient perceive the success of a root coverage procedure. The patient's satisfaction with the aesthetic outcome did not always match the professional scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo VO Fernandes, PhD, Study Director — A.T. Still University
Locations (1):
- Universidade Católica Portuguesa, Viseu, Viseu District, Portugal